CLINICAL TRIAL: NCT06226610
Title: A Phase 2 Double-Blind, Randomized, Placebo-Controlled Study to Assess the Efficacy of Dupixent in Adults With Refractory Post-Burn Pruritus in an Ambulatory Clinic
Brief Title: Dupixent in Adults With Refractory Post-Burn Pruritus in an Ambulatory Clinic
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-002
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-12

CONDITIONS: Pruritis
Keywords: Itching, itch
MeSH Terms: conditions — Pruritus | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: This is a dual-arm, two-site, randomized, placebo-controlled interventional Phase 2 randomized controlled clinical trial to estimate the potential effect size of Dupixent on improving post-burn pruritus symptoms. N=46 participants will be enrolled at a 1:1 intervention:control ratio.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study sponsor will supply all study drug (including placebo) as blinded kits. Study staff, investigators, and participants will be blinded to which treatment condition a participant has been randomized to. Note that the drug manufacturer will email codes to the pharmacists (who are unblinded) identifying the appropriate study drug for a particular participant. It is possible that participants may become unblinded to the obvious physical effects related to receiving Dupixent or placebo (pruritus improves or does not improve). Study staff will not discuss or speculate potential treatment arm allocation with participants based on participants' comments, questions, daily itch diary data, or physical observation. Study staff will encourage participants expressing resentful demoralization to remain in the study through their final visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARM 1 - Dupixent (Active Comparator): Two subcutaneous injection of 300mg Dupixent at visit 1 and every two weeks (+/- 2 days) for a total of 6 administrations. Injections may be administered in the thigh, lower abdomen or upper arm. The initial dose (two 300 mg doses) will be given in two different injection sites. There are not restriction or guidance regarding dose administration related to meals. No dose modifications will occur during study participation.
  Interventions: Drug: Dupilumab
- ARM 2 - Placebo (Placebo Comparator): Two subcutaneous injection of the placebo at visit 1 and every two weeks (+/- 2 days) for a total of 6 administrations. Injections may be administered in the thigh, lower abdomen or upper arm. The initial dose (two doses) will be given in two different injection sites. There are not restriction or guidance regarding dose administration related to meals. No dose modifications will occur during study participation.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dupilumab — injection every two weeks while on study
  Arms: ARM 1 - Dupixent
Other: Placebo — injection every two weeks while on study
  Arms: ARM 2 - Placebo

SUMMARY:
The goal of this study is to test the efficacy of Dupixent in improving post-burn itching symptoms versus the current standard of care.

DETAILED DESCRIPTION:
Participants will receive six injections of Dupixent or placebo (two 300 mg loading doses and one 300 mg dose every two weeks after that).

In addition, participants will be asked to complete questionnaires to determine daily itch severity, quality of life, treatment benefit, physical functioning, and pain interference.

Individual participants will require 13 weeks to complete all study visits.

ELIGIBILITY:
Inclusion Criteria:

• Persons 18-60 year old with post-burn hypertrophic scars of any size which required grafting or epidermal autografting for an acute burn injury, with continued complaint of pruritus due to inadequate relief from standard of care (medical management by antihistamine and neuroleptic medications) after at least four weeks and are a minimum of four weeks after their last grafting surgery, and who speak English sufficient to participate in the study.

Exclusion Criteria:

* Currently taking Dupixent for any other diagnosis
* known allergy to Dupixent
* pregnant and or lactating mothers
* anyone treated for pruritus using laser therapy
* currently receiving adequate relief for pruritis under standard of care medical management by antihistamine or neuroleptic medications
* Currently taking steroids
* persons with developmental delays or otherwise unable to complete measures
* prisoners or anyone otherwise unable to give their own consent or who is not their own guardian
* one or more of the following existing disorders: conjunctivitis; any co-existing dermatological condition except burns; any type of cancer; requiring dialysis; chronic Stage 3 or higher kidney disease; biliary disorder; gall bladder disorder; or another renal or hepatic disorder which, in the opinion of study physician, deems this study inappropriate for an eligible individual.
* Persons unable to provide their own consent, including prisoners when their incarcerated status is not itself the focus of study, are routinely excluded from clinical trials at this site
* We further exclude persons with other dermatological conditions (other than burn) , which may have pruritis or pain associated with them and who may be treated with medications other than Dupixent, and whose perceived benefit could confound our results.
* We similarly exclude anyone treated for pruritis by laser therapy as their perceived benefit could confound our results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Itch Severity Scale (ISS) Scores | 12 WEEKS
  Participants' Itch Severity Scale (ISS) scores will decrease more than 2.0 points after 12 weeks following initiating use of Dupixent

CONTACTS AND LOCATIONS:
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No